CLINICAL TRIAL: NCT01557959
Title: Phase II Study of Sequential Dose-Dense Chemotherapy and Dose-Intense Erlotinib for the Initial Treatment of Advanced Non-Small Cell Lung Cancer
Brief Title: Docetaxel, Cisplatin, Pegfilgrastim, and Erlotinib Hydrochloride in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU 62107; NCI-2009-01252 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00723138 (obsolete NCT alias)
Record Dates: First submitted 2012-02-14; First posted 2012-03-20 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; pegfilgrastim; Erlotinib Hydrochloride; Amplified Fragment Length Polymorphism Analysis; Pharmacogenomic Testing; Genetic Linkage; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemo, chemoprotection, antiangiogenesis therapy) (Experimental): Patients receive docetaxel IV over 1 hour on day 1, cisplatin IV over 1 hour on day 1, and pegfilgrastim subcutaneously on day 2. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after completion of docetaxel, cisplatin, and pegfilgrastim, patients receive oral erlotinib hydrochloride once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Biological: pegfilgrastim; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Genetic: polymorphism analysis; Other: pharmacogenomic studies; Genetic: genetic linkage analysis; Drug: docetaxel

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Optional correlative study
Genetic: polymorphism analysis — Correlative study
Other: pharmacogenomic studies — Correlative study
  Other Names: Pharmacogenomic Study
Genetic: genetic linkage analysis — Correlative study
  Other Names: linkage analysis
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT

SUMMARY:
This phase II trial is studying how well docetaxel given together with cisplatin and pegfilgrastim followed by erlotinib hydrochloride works in treating patients with stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving dose-dense combination chemotherapy together with pegfilgrastim and erlotinib hydrochloride may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if this regimen improves the time-to-progression for patients with advanced non-small cell lung cancer (NSCLC) compared to historical controls.

SECONDARY OBJECTIVES:

I. To assess response rate and median survival. II. To evaluate tumor biomarkers that could predict response and survival for patients treated with this regimen including endothelial growth factor receptor (EGFR) expression, EGFR Fluorescence in situ hybridization (FISH), and k-ras mutations.

III. To evaluate genetic polymorphisms as markers of response and survival for patients treated with this regimen including polymorphisms in XPD, XRCC1, XRCC3, and cyclin D1.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 1 hour on day 1, cisplatin IV over 1 hour on day 1, and pegfilgrastim subcutaneously (SC) on day 2. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after completion of docetaxel, cisplatin, and pegfilgrastim, patients receive erlotinib hydrochloride orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Documentation: Either histologic or cytologic documentation of non-small cell carcinoma (NSCLC) is necessary, and the following diagnostic categories are acceptable: squamous carcinoma, basaloid carcinoma, adenocarcinoma, bronchioloalveolar carcinoma, adenosquamous carcinoma, large cell carcinoma (not neuroendocrine), sarcomatoid carcinoma, and non-small cell carcinoma not otherwise specified (NOS); histologic or cytologic documentation of recurrence is required in patients who were previously completely resected
* Advanced Disease: Stage IIIB because of malignant pleural or pericardial effusion or stage IV disease
* Patients must be ineligible for Avastin or decline treatment with Avastin
* Prior Treatment: No prior chemotherapy or treatment with an EGFR inhibitor is allowed; brain metastasis must be under control (patient neurologically stable)
* All Patients must have Measurable or Non-Measurable Disease: measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension; the longest diameter of measurable lesions must be >= 20 mm with conventional techniques or >= 10 mm with spiral computed tomography (CT) scan; non-measurable disease includes the following:

  * Bone lesions
  * Brain metastasis or leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Tumor lesions situated in a previously irradiated area

    * Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
    * Granulocytes >= 1,500/ul
    * Platelets >= 100,000/ul
    * Creatinine =< upper limit of normal (ULN)
    * Bilirubin =< 1.5 mg/dl
    * Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 1.5 x ULN
    * Alkaline (Alk.) phosphatase (phos.) =< 2.5 x ULN
* Patients must provide verbal and written informed consent to participate in the study

Exclusion Criteria:

* Patients who are pregnant or nursing because of significant risk to the fetus/infant
* Patients with neuropathy >= grade 2
* Patients with a psychiatric illness which would prevent the patient from giving informed consent
* Patients who are unable to take oral medications
* Women with child-bearing potential or men who are sexual partners of women with child-bearing potential who are not willing to practice adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Petty, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Petty WJ, Laudadio J, Brautnick L, Lovato J, Dotson T, Streer NP, Weaver KE, Miller AA. Phase II trial of dose-dense chemotherapy followed by dose-intense erlotinib for patients with newly diagnosed metastatic non-small cell lung cancer. Int J Oncol. 2013 Dec;43(6):2057-63. doi: 10.3892/ijo.2013.2122. Epub 2013 Oct 3. PMID 24100924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy)
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy)
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Determined using RECIST. Estimated using the Kaplan-Meier method. Log-rank tests will be used to test for differences and Cox proportional hazards regression modeling will be used to adjust for patient demographics and characteristics such as smoking status at baseline (actively/non-actively smoking). Progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy)
Number analyzed (Participants) | 45
months | 4.63 [3.68 to 6.05]

2. Secondary Outcome: Response Rate Among Subgroups of Patients According to Molecular Profiles Including Tumor Characteristics and Genetic Polymorphisms From Peripheral Blood
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Pre-specified that data is only presented for the subgroups "Low Cyclin D1" and "High Cyclin D1".
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Cyclin D1 | High Cyclin D1
Number analyzed (Participants) | 16 | 15
Participants
  Progressive disease | 3 | 4
  Stable disease | 9 | 9
  Partial response | 4 | 2

3. Secondary Outcome: Median Survival Among Subgroups of Patients According to Molecular Profiles Including Tumor Characteristics and Genetic Polymorphisms From Peripheral Blood
Time Frame: 2 years
Measure: Median (Standard Error); unit: Months
Arm/Group | Low Cyclin D1 | High Cyclin D1
Number analyzed (Participants) | 16 | 15
Months | 20.5 (7.7) | 8.0 (10.7)

ADVERSE EVENTS:
Description: 44 of the 45 patients had completed therapy at the time of reporting. Adverse events reflect those 44 patients.
Arm/Group | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy)
Serious Adverse Events (participants affected / at risk) | 39/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy) (N=44)
Low WBC (Investigations) | 3 (3)
low Platelets (Investigations) | 3 (3)
Low Hemoglobin (Investigations) | 8 (8)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Anorexia (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1)
Low ANC (Investigations) | 7 (7)
Dizziness (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Weight loss (General disorders) | 1 (1)
hyperglycemia (Investigations) | 3 (3)
hypocalcemia (Investigations) | 7 (7)
hypomagnesemia (Investigations) | 2 (2)
hyponatremia (Investigations) | 5 (5)
hypokalemia (Investigations) | 7 (7)
hypoalbuminemia (Investigations) | 4 (4)
serum glutamic pyruvic transaminase (Investigations) | 2 (2)
hypophosphatemia (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 5 (5)
serum glutamic oxaloacetic transaminase (Investigations) | 2 (2)
hyperkalemia (Investigations) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Dysphagia (General disorders) | 1 (1)
Fever without neutropenia (General disorders) | 1 (1)
Urinary frequency/urgency (General disorders) | 1 (1)
Edema: limb (Vascular disorders) | 1 (1)
Hypoxia (Investigations) | 5 (5)
Dehydration (General disorders) | 3 (3)
Confusion (General disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7)
Acidosis (Investigations) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Partial Thromboplastin Time (Investigations) | 2 (2)
Pain: Joint (General disorders) | 1 (1)
Arthritis (non-septic) (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pain: Bone (General disorders) | 1 (1)
Pain: Chest wall (General disorders) | 2 (2)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 1 (1)
"Hemorrhage, GI: Duodenum" (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage Stomach (Vascular disorders) | 1 (1)
"Hemorrhage, CNS" (Blood and lymphatic system disorders) | 1 (1)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Flu-like syndrome (Infections and infestations) | 1 (1)
Lymphopenia (Investigations) | 12 (12)
Muscle weakness (General disorders) | 2 (2)
Nail changes (General disorders) | 1 (1)
"Stricture/stenosis (including anastomotic), GI: Esophagus" (General disorders) | 1 (1)
Pain: Extremity-limb (General disorders) | 1 (1)
Pain (unspecified) (General disorders) | 1 (1)
Pain: Pleura (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 6 (6)
"Hemorrhage, GI: Rectum" (Blood and lymphatic system disorders) | 1 (1)
"Hemorrhage, pulmonary/upper respiratory: Respiratory tract NOS" (Blood and lymphatic system disorders) | 1 (1)
Infection with unknown ANC: Blood (Infections and infestations) | 1 (1)
Syncope (fainting) (General disorders) | 3 (3)
Vasovagal episode (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Urinary with low grade neutropenia (Infections and infestations) | 1 (1)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Pain: Tumor pain (General disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils: Conjunctiva (Infections and infestations) | 1 (1)
"Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided" (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: External ear (General disorders) | 1 (1)
Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Blood Infection with high grade neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemo, Chemoprotection, Antiangiogenesis Therapy) (N=44)
Low WBC (Investigations) | 41 (41)
low Platelets (Investigations) | 41 (41)
Low Hemoglobin (Investigations) | 36 (36)
Nausea (Gastrointestinal disorders) | 43 (43)
Vomiting (Gastrointestinal disorders) | 41 (41)
Diarrhea (Gastrointestinal disorders) | 37 (37)
Anorexia (General disorders) | 38 (38)
Alkaline phosphatase (Investigations) | 44 (44)
Creatinine (Investigations) | 44 (44)
Proteinuria (Investigations) | 7 (7)
Hair loss (General disorders) | 12 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (21)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 44 (44)
Hypertension (General disorders) | 4 (4)
Hypotension (Cardiac disorders) | 9 (9)
Neuropathy: sensory (Cardiac disorders) | 12 (14)
Neuropathy: motor (Nervous system disorders) | 4 (4)
Low ANC (Investigations) | 37 (37)
Pain (unspecified) (General disorders) | 44 (44)
Dizziness (General disorders) | 10 (10)
Taste alteration (General disorders) | 7 (7)
Insomnia (General disorders) | 7 (7)
Neurology (Nervous system disorders) | 44 (44)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 44 (45)
Rigors/chills (General disorders) | 44 (44)
Sweating (General disorders) | 2 (2)
Fatigue (General disorders) | 41 (41)
Weight loss (General disorders) | 8 (8)
hyperglycemia (Investigations) | 28 (28)
hypoglycemia (Investigations) | 4 (4)
hypercalcemia (Investigations) | 44 (44)
hypocalcemia (Investigations) | 37 (37)
hypomagnesemia (Investigations) | 17 (17)
hyponatremia (Investigations) | 39 (39)
hypokalemia (Investigations) | 36 (36)
Bicarbonate serum-low (Investigations) | 44 (44)
hypoalbuminemia (Investigations) | 40 (40)
hyperbilirubinemia (Investigations) | 44 (44)
serum glutamic pyruvic transaminase (Investigations) | 10 (10)
hypophosphatemia (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 43 (43)
Pain: Head/headache (General disorders) | 9 (9)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
serum glutamic oxaloacetic transaminase (Investigations) | 42 (42)
hyperkalemia (Investigations) | 43 (43)
hypernatremia (Investigations) | 44 (44)
Phlebitis (Vascular disorders) | 3 (3)
Ocular/Visual - Other (Eye disorders) | 3 (3)
Dysphagia (General disorders) | 3 (3)
Fever without neutropenia (General disorders) | 43 (43)
Cardiac (Cardiac disorders) | 44 (44)
Infection - Other (Infections and infestations) | 44 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (27)
Auditory/Ear (Ear and labyrinth disorders) | 44 (44)
Edema: head and neck (Vascular disorders) | 2 (2)
Edema: limb (Vascular disorders) | 10 (12)
Edema: trunk/genital (General disorders) | 3 (3)
Heartburn/dyspepsia (General disorders) | 6 (6)
Dry mouth (General disorders) | 2 (2)
Dehydration (General disorders) | 7 (7)
Confusion (General disorders) | 4 (4)
Pruritus/itching (General disorders) | 9 (9)
Mood alteration: Agitation (General disorders) | 3 (3)
Anxiety (General disorders) | 6 (6)
Depression (General disorders) | 6 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (8)
Pain: Abdomen (General disorders) | 7 (7)
Acidosis (Investigations) | 3 (3)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 9 (9)
Partial Thromboplastin Time (Investigations) | 4 (4)
Alkalosis (Investigations) | 2 (2)
Pain: Joint (General disorders) | 11 (13)
Arthritis (non-septic) (General disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pain: Back (General disorders) | 9 (9)
Pain: Bone (General disorders) | 10 (12)
Infection with normal ANC or Grade 1 or 2 neutrophils: Bronchus (Infections and infestations) | 3 (3)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pain: Chest/thorax (General disorders) | 3 (3)
Pain: Chest wall (General disorders) | 4 (4)
Seizure (Nervous system disorders) | 2 (2)
Dry eye syndrome (Eye disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15)
Hemorrhage respiratory (Vascular disorders) | 8 (8)
Neuropathy: cranial: CN VII Motor-face; Sensory-taste (General disorders) | 2 (2)
Glomerular filtration rate (Investigations) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 42 (42)
"Watery eye (epiphora, tearing)" (Eye disorders) | 3 (3)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (4)
Lymphopenia (Investigations) | 19 (19)
Memory impairment (General disorders) | 2 (2)
Hemorrhage GI: Oral cavity (Vascular disorders) | 2 (2)
Muscle weakness (General disorders) | 9 (9)
Pain: Muscle (General disorders) | 8 (8)
Nail changes (General disorders) | 7 (7)
Pain: Extremity-limb (General disorders) | 3 (3)
Palpitations (General disorders) | 2 (2)
Pain: Throat/pharynx/larynx (General disorders) | 2 (2)
Pain: Pleura (General disorders) | 8 (8)
Lung infection (Infections and infestations) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash: dermatitis associated with radiation: Chemoradiation (Skin and subcutaneous tissue disorders) | 2 (2)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 8 (8)
Sinus tachycardia (Cardiac disorders) | 9 (9)
Infection with normal ANC or Grade 1 or 2 neutrophils: Skin (cellulitis) (Infections and infestations) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils: Vagina (Infections and infestations) | 2 (2)
blurred vision (Eye disorders) | 2 (2)
Pain: Buttock (General disorders) | 2 (2)
Pain: Tumor pain (General disorders) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils: Nose (Injury, poisoning and procedural complications) | 2 (2)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 44 (44)
Hemorrhage pulmonary/upper respiratory (Vascular disorders) | 6 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils: Conjunctiva (Infections and infestations) | 2 (2)
"Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower" (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuropathy: cranial: CN VIII Hearing and balance (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes